CLINICAL TRIAL: NCT06349655
Title: Real-World Effectiveness and Safety of Oral Azvudine in Hospitalized Patients With COVID-19: A Multicenter, Retrospective, Cohort Study
Brief Title: The Real-world Clinical Study of Azvudine Tablets in the Treatment of COVID-19
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Zhengzhou University (Other)
Collaborators: Henan Provincial Chest Hospital (Other); The Affiliated Infectious Disease Hospital of Zhengzhou University (Unknown); The Fifth People's Hospital of Anyang (Unknown); Shangqiu Municipal Hospital (Unknown); Nanyang Central Hospital (Other); Luoyang Central Hospital (Other); Guangshan County People's Hospital (Unknown); Fengqiu County People's Hospital (Unknown)
Responsible Party: Principal Investigator, Zhigang Ren, Professor, The First Affiliated Hospital of Zhengzhou University
Other Study IDs: 2023-KY-0865-001
Record Dates: First submitted 2024-04-02; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COVID-19; Azvudine
MeSH Terms: conditions — COVID-19 | interventions — azvudine; nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Azvudine: COVID-19 patients with Azvudine treatment
  Interventions: Drug: Azvudine
- Paxlovid: COVID-19 patients with Paxlovid treatment
  Interventions: Drug: Paxlovid
- Control: COVID-19 Patients who have not been treated with Azvudine or Paxlovid

INTERVENTIONS:
Drug: Azvudine — Antiviral drug
  Groups: Azvudine
Drug: Paxlovid — Antiviral drug
  Other Names: Nirmatrelvir/Ritonavir
  Groups: Paxlovid

SUMMARY:
To establish a real-world clinical cohort and database of Azvudine in the treatment of SARS-CoV-2 infection, and to provide stable and reliable evidence for the clinical efficacy and safety evaluation of azvudine in the treatment of SARS-CoV-2 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years old (including the cut-off value), regardless of gender;
2. Patients diagnosed with 2019-ncov infection according to the diagnostic criteria of the latest edition of the Diagnosis and Treatment Plan for 2019-ncov Pneumonia issued by the Health Commission of China;
3. Informed consent has been signed.

Exclusion Criteria:

1. Known or suspected allergic to the components of Azivudine tablets;
2. Patients with severe liver, kidney, heart and other organ damage;
3. Pregnant or lactating women who planned to give birth during or within 6 months after the trial;
4. Had participated in other clinical trials or were using investigational drugs within 12 weeks before medication;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People who have COVID-19 and have an indication for Azvudine or Paxlovid.
Sampling Method: Non-Probability Sample
Enrollment: 32864 (Actual)
Dates: Start 2023-12-05 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
All-cause death | Up to 30 days (form the date of confirmed COVID-19)
  All-cause death was ascertained by electronic medical records.

SECONDARY OUTCOMES:
Composite disease progression | Up to 30 days (form the date of confirmed COVID-19)
  Disease progression is defined as the occurrence of death, progression to severe or critical disease in mild or moderate patients, and the occurrence of death, progression to critical disease in severe patients. Severe disease is defined as respiratory rate ≥ 30 times/minute, or resting oxygen saturation ≤ 93%, or PaO2/FiO2 ≤ 300 mmHg, or lung lesions progressing >50% at 24-48 hours. Critical disease is defined as the need for mechanical ventilation, or shock, or ICU monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Zujiang Yu, Dr., Study Director — The First Affiliated Hospital of Zhengzhou University
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wang F, Jia B, Li G, Jin X, Yang M, Li G, Zhang S, Qian G, Luo H, Cheng M, Wang L, Zhang D, Li S, Liang H, Ren Z. Real-world effectiveness and safety of oral azvudine versus Paxlovid in patients with COVID-19 and pre-existing hypertension: a multicentre, retrospective, cohort study in Henan Province, China. BMJ Open. 2025 Jun 27;15(6):e090230. doi: 10.1136/bmjopen-2024-090230. PMID 40578868
- [Derived] Su G, Gao F, Yang M, Wang L, Liang L, Li S, Li G, Han N, Li G, Qian G, Zhang S, Luo H, Zhang D, Liang H, Ren Z. Effectiveness of azvudine versus nirmatrelvir/ritonavir for hospitalized patients with SARS-CoV-2 infection and pre-existing liver diseases. Virol J. 2025 May 19;22(1):147. doi: 10.1186/s12985-025-02771-1. PMID 40389963